CLINICAL TRIAL: NCT03275142
Title: Icare Tonometry Effects on Keratometry Readings, Topography Readings, and Corneal Staining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comprehensive EyeCare of Central Ohio (Other)
Collaborators: Icare USA (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 170608-1
Record Dates: First submitted 2017-07-26; First posted 2017-09-07 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Evaluation of Corneal Stability Post-applanation
MeSH Terms: interventions — Manometry

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Only the Investigator will be interpreting outcomes. The technician/care provider will perform all testing and will mask the investigator to which eye tonometry was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Icare Applanation (Experimental): Evaluation of corneal stability post-applanation with Icare tonometer via pre and post applanation keratometry readings with IOL Master, topography with Pentacam, fluorescein corneal staining. Patient's OD and OS are randomized into "study" or control, then undergo applanation with Icare. Investigator is masked as to which eye has undergone applanation.
  Interventions: Device: Icare tonometer
- No ICare Applanation (Active Comparator): Evaluation of corneal stability post-applanation with Icare tonometer via pre and post applanation keratometry readings with IOL Master, topography with Pentacam, fluorescein corneal staining. Patient's OD and OS are randomized into "study" or control, then undergo applanation with Icare. Investigator is masked as to which eye has undergone applanation.
  Interventions: Device: Icare tonometer

INTERVENTIONS:
Device: Icare tonometer — Icare tonometry effects of keratometry readings, topography, and corneal staining to demonstrate that the Icare tonometer does not alter subsequent evaluation or testing. This would allow IOP testing to be performed by technical staff at any time during the examination process without affecting subsequent tests. A total of fifteen patients at each of four sites will be evaluated using Icare tonometers provided by Icare USA. The investigator will be masked as to which eye will undergo Icare tonometry. Both the study eye and the control eye will undergo pre-tonometry and post-tonometry testing; Keratometry readings, IOL master, Topography via Pentacam, and corneal staining with fluorescein using the Oxford scoring scale.
  Other Names: Icare; applanation; tonometry

SUMMARY:
To demonstrate that the Icare tonometer does not alter Keratometry readings, topography, or corneal staining. This would therefore allow intraocular pressure (IOP) testing to be done at any time during an exam, without affecting other testing. This may improve office-flow and spare patients from returning for another exam for additional testing.

DETAILED DESCRIPTION:
Four sites will enroll fifteen subjects each. Individual sites will identify their patients using numbers 1-15. The link to their identity will be stored in their records but will not be forwarded to other investigators. Only the originating site will have the identity log linking the participants to the study records. All patients over age 18 in the patient clinic are eligible for inclusion. Staff members and employees may also participate. Following informed consent, each patient will undergo visual acuity testing, keratometry readings by IOL Master, topography testing by Pentacam, and corneal staining evaluation with fluorescein using the Oxford scoring scale on both eyes. Once all three tests are completed, the Icare tonometer will be used to check the intraocular pressure (IOP) on one eye only. The investigator will be masked as to which eye will undergo applanation. Immediately following the IOP check, corneal staining, topography and keratometry readings will be repeated. The unchecked eye will serve as a control as there may be mild variations in topography or IOL Master even without applanation. Following the repeated testing, the control eye will also undergo applanation to document IOP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Demonstration of corneal stability post-applanation with the Icare tonometer. | 30 minutes
  Demonstration that the Icare tonometer does not alter keratometry readings performed by IOL Master, topography performed by Pentacam HR, or corneal staining as evaluated at slit-lamp with fluorescence as compared to the Oxford Grading Scale

SECONDARY OUTCOMES:
Average keratometric measurement differences pre and post- tonometry with ICare Tonometer. | 10 minutes
  Evaluation of average keratometric difference pre and post-tonometry with ICare via Pentacam HR and IOL Master.
Total cylinder differences pre and post-tonometry with ICare tonometer. | 10 minutes
  Total cylinder differences pre and post-tonometry with ICare Tonometer via Pentacam HR and IOL Master.
Difference in corneal staining pre and post-tonometry with ICare Tonometer. | 10 minutes
  Difference in corneal staining pre and post-tonometry with ICare Tonometer as compared to the Oxford Scoring Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Beckman, M.D., Study Director — Comprehensive EyeCare of Central Ohio
Locations (1):
- Comprehensive EyeCare of Central Ohio, Westerville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Only the originating site of study will have the identity log linking the participants to the study records.

DOCUMENTS (2):
  • Informed Consent Form (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT03275142/ICF_000.pdf
  • Study Protocol (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT03275142/Prot_001.pdf